CLINICAL TRIAL: NCT04747132
Title: Effectiveness of a Telegeriatric Intervention in Older Adults During the Covid-19 Contingency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Iberoamericana A.C., Mexico (Other)
Responsible Party: Principal Investigator, Oscar Rosas Carrasco, Investigator, Universidad Iberoamericana A.C., Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SALUD-2021-Telegeria
Record Dates: First submitted 2021-02-06; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Effectiveness
Keywords: Aged; Internet-Based Intervention; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individualized geriatric medical counseling, psychological counseling, nutritional counseling and physical activity counseling through the internet
  Interventions: Other: Telegeriatric intervention
- Control group (No Intervention): Health guidance through standardized audiovisual educational material through Intenert

INTERVENTIONS:
Other: Telegeriatric intervention — Individualized, comprehensive and specialized counseling for older adults through the Internet
  Other Names: Telenutrition intervention
  Arms: Intervention group

SUMMARY:
The purpose of this studdy is to assess the effectiveness of a telegeriatric intervention

DETAILED DESCRIPTION:
The patients were recruited from a cohort study in which the participants had previously signed an informed consent in which they allowed contact to participate in new studies, participants who met the inclusion criteria in the original database were recruited and signed an electronic informed consent of the new study. A comprehensive geriatric assessment was generated to assess whether they were candidates even due to changes in health status that could change over time since their last assessment, they were recruited until the expected sample size was obtained, and they were randomized, blinding the participants to belong to the intervention group (individualized care: geriatrics, psychology, physical activity and nutrition) or the control group (orientation in standardized health issues through audiovisual educational material)

ELIGIBILITY:
Inclusion Criteria:

* Adults 60 years and over
* Who agree to participate in the study.

Exclusion Criteria:

* Older adults who are in a systematic exercise program or directed food restriction programs
* Physical, sensory or cognitive disabilities that prevent exercise, includes Mini Mental State Examination less than 20 points of the total score
* Any condition acute or chronic health conditions that clinical staff judge as an impediment to the exercise program or remote monitoring
* Recent major or limb surgery
* Orthopedic conditions that would impede the exercise program
* Any problem swallowing
* Previous mental disorders such as disorder and schizophrenia
* Not having personal access to the WhatsApp application via video call.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Visual analog scale of the European quality of life questionnaire | Change from baseline to week 12
  The visual analog scale of the European quality of life questionnaire, adapted and validated to Spanish, Mexico (EQ5D-VAS) will be used. Which consists of a visual analog scale, its total score ranges from 0 to 100 points, the higher the score, the better the quality of life, it will be considered as a continuous quantitative variable. (Juárez-Cedillo T et al., 2015) Change from baseline to week 12
Physical performance. | Change from baseline to week 12
  It will be evaluated through the short physical performance test (SPPB), which is a test that includes three dimensions: strength. March and balance, your score ranges from 0 to 12 points, the higher the score the better the physical performance, it will be considered as a continuous quantitative variable. (Guralnik JM et al., 1989) Change from baseline to week 12
Depressive symptoms | Change from baseline to week 12
  It will be evaluated using the CESD scale 7 items validated into Spanish in Mexico. His score ranges from 0 to 21 points, the higher the score, the greater the depressive symptoms. The total score will be considered as a continuous quantitative variable. (Salinas-Rodríguez A et al., 2014) Change from baseline to week 12
Symptoms of anxiety. | Change from baseline to week 12
  It will be evaluated through the geriatric anxiety inventory, which is validated in Spanish, consists of 20 dichotomous items, its total score ranges from 0 to 20, the higher the score, the greater the anxiety symptoms. It will be considered as a continuous quantitative variable. (Márquez-González M et al., 2012) Change from baseline to week 12
Body composition | Change from baseline to week 12
  It will be evaluated by using the OMROM HBF-514C® 50 Hz portable electrical bioimpedance bascule Change from baseline to week 12
Anthropometric measures | Change from baseline to week 12
  It will be evaluated by using the SECA anthropometric tape Change from baseline to week 12
Dietary intake | Change from baseline to week 12
  It will be evaluated by using the ASA24 software for 24-hour reminder collection by multiple steps.
  Change from baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Rosas Carrasco, Principal Investigator — Universidad Iberoamericana
Locations (1):
- Universidad Iberoamericana, Mexico City, Mexico City, Mexico